CLINICAL TRIAL: NCT01969461
Title: Comparing the Effectiveness of Two Alcohol+Adherence Interventions for HIV+ Youth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wayne State University (Other)
Collaborators: Westat (Other); City University of New York, School of Public Health (Other); University of California, San Diego (Other); Medical University of South Carolina (Other); University of California, Los Angeles (Other); Columbia University (Other); University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Sylvie Naar-King, Professor, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1R01AA022891-01 (NIH)
Record Dates: First submitted 2013-10-17; First posted 2013-10-25 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2017-01

CONDITIONS: HIV
Keywords: HIV positive; Adolescents; Adolescent Trials Network; Comparative Effectiveness Trial; Implementation; Adherence Intervention; Alcohol Intervention
MeSH Terms: conditions — HIV Seropositivity; Adherence Interventions | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Healthy Choices: MET CHW Clinic (Experimental): The 4-session Motivational Enhancement Therapy (MET) intervention will address alcohol use and HIV medication (ART) adherence. Sessions will be delivered in the CLINIC by a CHW (outreach worker, etc) already providing services in the clinic. The intervention is based on Motivational Interviewing (MI) techniques, building motivation for change by eliciting and reinforcing change talk.
  Interventions: Behavioral: Motivational Enhancement Therapy (MET)
- Healthy Choices: MET CHW Home (Active Comparator): The 4-session Motivational Enhancement Therapy (MET) intervention will address alcohol use and HIV medication (ART) adherence. Sessions will be delivered in the HOME by a CHW (outreach worker, etc) already providing services in the clinic. The intervention is based on Motivational Interviewing (MI) techniques, building motivation for change by eliciting and reinforcing change talk.
  Interventions: Behavioral: Motivational Enhancement Therapy (MET)

INTERVENTIONS:
Behavioral: Motivational Enhancement Therapy (MET) — The 4-session MET intervention will address alcohol use and HIV medication (ART) adherence. Sessions will be delivered in the clinic or the home by a CHW (outreach worker, etc) already providing services in the clinic. In sessions 1 and 2 (each behavior will get its own session), CHW will elicit the client's view of the problem using MI techniques, building motivation for change by eliciting and reinforcing change talk. The CHW will deliver feedback and discuss the consideration of a behavior change plan option, and the client sets the change plan goal and consolidates commitment. In the last two sessions, the CHW will review the change plan, continue to elicit and reinforce change talk, problem-solve barriers, consolidate commitment, and consider strategies to maintain behavior change.
  Other Names: Motivational Interviewing

SUMMARY:
Alcohol use among persons with HIV exacerbates health problems and accelerates HIV disease progression. Antiretroviral therapy (ART) is the single most important treatment for people living with HIV. However, ART adherence is suboptimal among adolescents and young adults living with HIV, the age group with the fastest growing rates of HIV infection, and great risk of engaging in risky behaviors such as alcohol use. The proposed study will compare the effectiveness of home-based versus clinic-based "Healthy Choices", a brief, 4- session intervention using Motivational Enhancement Therapy (MET) to address alcohol use, medication adherence, and health outcomes in youth living with HIV (YLH) using a repeated measures design. Unlike previous trials, Healthy Choices will be tested in a "real world" clinical setting and be delivered by community health workers (CHW: already members of the HIV care team). The study population will consist of YLH, ages 16-24, who are current patients at 5 ATN sites. Site staff will recruit potential participants. Youth will be randomized to receive Healthy Choices, either clinic-based or home-based delivered by the same CHW in both conditions. Outcomes are measured at baseline, 4-, 7-, and 13-months. Data collection for biological measures will be through medical record extraction, and self-reported measures will occur using a brief Web-based CASI (computer-administered self-interviewing) survey on an iPad. All intervention sessions will be audio-recorded for MITI fidelity coding, and investigators will support local supervisors during the active intervention phase. We will conduct qualitative interviews with CHWs, supervisors and organization leaders at the end of the trial to obtain information about barriers and facilitators of implementation. Thus, the proposed trial will allow us to use a Type 1 Effectiveness-implementation hybrid design to pilot a sustainable model of MI implementation in real-world youth care settings towards the goals of 1) examining the effectiveness, cost-effectiveness, and scalability of an efficacious behavioral intervention when delivered by CHWs in real-world adolescent HIV care settings; 2) gathering information about who responds under what contexts; and 3) increasing our understanding of the barriers and facilitators for future implementation. The primary hypothesis is that YLH receiving home-based MET will have greater improvements in alcohol use and viral load than YLH receiving clinic-based MET.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected
* Ability to speak and understand English
* Prescribed antiretroviral therapy
* Detectable viral load in the last month

Exclusion Criteria:

* Not fluent in English
* History of sever learning disability, mental retardation, major psychiatric disorders (e.g., schizophrenia, bipolar disorder, major depression with psychotic features, etc).
* Participation in another adherence intervention trial
* On ART due to pregnancy

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 400 (Estimated)
Dates: Start 2014-07; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change in Alcohol Use from Baseline to 9 months post intervention | Baseline, 4-, 7-, and 13-months
  We will use multiple methods of assessing use including calendar-based interview, biomarker, and self-report questionnaire.
Change in Viral Load from Baseline to 9 months post intervention | Baseline, 4-, 7-, and 13-months
  Viral load will be extracted from medical records, though we have budgeted to collect a percentage of viral loads for youth who drop out of care or transfer to a care setting where records are not available.

SECONDARY OUTCOMES:
Change in Medication Adherence from Baseline to 9 months post intervention | Baseline, 4-, 7-, and 13-months
  We will use self-report and interviews that have been successful in our previous trials.
Change in Sexual Risk from Baseline to 9 months post intervention | Baseline, 4-, 7-, and 13-months
  We will use self-report and interviews that have been successful in our previous trials.
Change in Other Substance Use (not alcohol use) from Baseline to 9 months post intervention | Baseline, 4-, 7-, and 13-months
  Objective measures are cost prohibitive (e.g., MEMS, hair assays, STI tests, urine screens) for these secondary outcomes; thus we will use self-report and interviews that have been successful in our previous trials.

OTHER OUTCOMES:
Barriers and Facilitators of the MI Implementation Process | 4 months post baseline
  The qualitative interview guide (with input from Dr. Norton, consultant) will focus on barriers and facilitators of implementation experienced at the individual, clinic, protocol team, and organizational level. Both positive and potentially negative outcomes will be elicited. Interviews will be conducted at the end of the MET intervention phase to assess sustainability.
Barriers and Facilitators of the MI Implementation Process | 13 months post Baseline
  The qualitative interview guide (with input from Dr. Norton, consultant) will focus on barriers and facilitators of implementation experienced at the individual, clinic, protocol team, and organizational level. Both positive and potentially negative outcomes will be elicited. Interviews will be conducted at the end of the trial to assess sustainability.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Naar-King, PhD, Principal Investigator — Wayne State University
Locations (1):
- Adolescent Trials Network (ATN) Sites, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Naar S, Robles G, MacDonell KK, Dinaj-Koci V, Simpson KN, Lam P, Parsons JT, Sizemore KM, Starks TJ. Comparative Effectiveness of Community-Based vs Clinic-Based Healthy Choices Motivational Intervention to Improve Health Behaviors Among Youth Living With HIV: A Randomized Clinical Trial. JAMA Netw Open. 2020 Aug 3;3(8):e2014650. doi: 10.1001/jamanetworkopen.2020.14650. PMID 32845328